CLINICAL TRIAL: NCT01434641
Title: Rapid Stress/Rest Single-Day Tc-99m Sestamibi Myocardial SPECT
Brief Title: Rapid Stress/Rest Single-Day Tc-99m Sestamibi Myocardial Single Photon Emission Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REGA-10K09
Record Dates: First submitted 2011-08-29; First posted 2011-09-15 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Disease
Keywords: myocardial perfusion SPECT; wide beam reconstruction; Tc-99m sestamibi
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- low-dose stress MPI SPECT (Other): Patients will receive a low-dose stress/high-dose rest protocol. Subject results are compared to archived patients undergoing a standard protocol./
  Interventions: Other: low-dose stress MPI SPECT

INTERVENTIONS:
Other: low-dose stress MPI SPECT — novel low-dose rest/high-dose Tc-99m sestamibi SPECT protocol with wide beam reconstruction SPECT processing

SUMMARY:
This protocol details a novel myocardial perfusion Single Photon Emission Computed Tomography (SPECT) protocol wherein patients receive a low-dose (6 mCi) of Tc-99m sestamibi during exercise or regadenoson pharmacologic stress and undergo a full-time SPECT acquisition processed with Wide Beam Reconstruction (WBR). Immediately thereafter patients receive a high-dose (30-35 mCi) of Tc-99m sestamibi at rest and undergo a half-time rest scan, also processed with WBR. All enrolled research subjects will undergo both the initial stress and subsequent rest scan.

The radiation exposure associated with this new stress/rest protocol is equivalent to that of the conventional rest/stress protocol presently in routine clinical uses at SLRHC.

Eventually, when and if this novel stress/rest protocol is adopted in routine clinical practice, patients with normal stress scans would receive only 6 mCi of Tc-99m sestamibi (331 mSv in men, 241 mSv in women) and spend only approximately one hour in the Nuclear Medicine Laboratory.

All patients presenting to the Nuclear Medicine Laboratory for evaluation of known or suspected coronary artery disease will be candidates for enrollment. Fifty patients undergoing treadmill exercise stress and 50 patients undergoing regadenoson pharmacologic stress will be enrolled. Pregnant and breast-feeding patients will not be eligible.

DETAILED DESCRIPTION:
Specific Aims:

To validate acceptable image quality and the stress/rest myocardial count density ratio (as defined below) of the Rapid Stress/Rest Protocol

Experimental Design and Methods:

Validation of the stress/rest myocardial count density ratio achieved using a standard rest/stress protocol incorporating a conventional 3:1 stress/rest Tc-99m radiopharmaceutical dose ratio.

Human subjects:

To determine the stress/rest myocardial count density ratio encountered using existing rest/stress imaging protocols in routine clinical practice, 100 consecutive patients undergoing either exercise or pharmacologic stress (dipyridamole or regadenoson) myocardial perfusion SPECT were included. The stress/rest Tc-99m sestamibi/Tc-99m tetrofosmin radiopharmaceutical dose ratio was 3:1 in all patients. Stress and rest maximal myocardial counts were determined from reconstructed tomograms using Evolution software (GE Healthcare).

The Investigational, novel stress/rest protocol:

Human Subjects: Characteristics and Plans for Recruitment 100 patients, who give their consent, presenting for myocardial perfusion SPECT in whom exercise or pharmacologic stress is clinically indicated will be enrolled prospectively. There will be no bias in selection of patients with regard to gender or racial/ethnic composition. 50 patients will be stressed with exercise. 50 additional patients will receive pharmacologic stress with the on-label dose of Regadenoson. All patients will receive the appropriate dose of radiotracer according to their size and weight. Pregnant women and those who are breast feeding will not be enrolled.

Patient Informed Consent:

Written informed consent will be obtained by either the Principal Investigator, the PI's research assistant (a physician), a Nuclear Medicine resident, or a Cardiology fellow (who will supervise and monitor the stress testing).

Methods - Imaging and Data Analysis:

The rapid stress/rest protocol, as described above, will be performed using the GE Ventri, MG or Maxxus dual-head supine scintillation camera and UltraSPECT Wide Beam Reconstruction (WBR) software. Both stress and rest SPECT will be performed in all patients, even if the initial stress images are normal.

Images will be interpreted and reported in the standard fashion for clinical patient management, characterizing perfusion defects in terms of location, extent, severity, reversibility, and function in terms of volume, regional wall motion and wall thickening.

Patient flow:

1. Upon arrival in the Nuclear Medicine Laboratory, patients will be interviewed regarding their medical history and a limited physical examination will be performed (as routinely performed for all clinically-indicated myocardial perfusion scans), and informed consent will be obtained for enrollment in this research study.
2. Patients able to perform treadmill exercise to 85% of their age-predicted maximum heart rate will undergo treadmill exercise stress. In the remainder of patients pharmacologic stress will be achieved with intravenous regadenoson. A stress dose of 5-7 mCi (adjusted for patient weight and chest circumference) Tc-99m sestamibi will be administered intravenously.
3. Post-stress gated SPECT will be acquired 30-60 min. thereafter using a full-time stress (12 min.) acquisition protocol, and processed using "half-time" Wide Beam Reconstruction software (i.e."half-dose" WBR protocol).
4. Within 60 minutes thereafter patients will receive an additional intravenous dose of 35-42 mCi (adjusted for patient weight and chest circumference) Tc-99m sestamibi at rest.
5. Resting gated SPECT will be acquired 40-60 minutes thereafter using a half-time resting (7.5 min.) acquisition protocol, and processed using "half-time" Wide Beam Reconstruction software (i.e. half-time" WBR protocol).
6. The estimated time for the entire study is approximately 3 hrs, which is slightly less than the time fro the standard rest/stress protocol the investigators now use.

Scans will be assessed for image quality using a 5-point subjective scale used in several reports the investigators have published previously (in references #2 and #3 below):

The image quality of the stress and rest perfusion tomograms and the gated tomograms is graded visually using a 5-point scale: 1 (poor) - 5 (excellent). Myocardial count density and uniformity, endocardial and epicardial edge definition, visualization and definition of the right ventricle, and background noise are parameters considered subjectively when grading image quality. In addition to those same attributes considered when grading the summed perfusion tomograms, the definition of the left ventricular cavity at end-systole and the temporal smoothness of the gated frames are also considered when grading the post-stress and rest gated images.

Stress and rest absolute myocardial count density and the stress:rest myocardial count density ratio will be determined from processed tomograms using General Electric Xeleris computer software. Count density is basically the "information density" of the scan. In general, as for all of nuclear imaging, the higher the count density, the better the image quality, the lower the incidence of scan artifacts, and the greater the clinical value of the scan.

The rest/stress myocardial count density ratio achieved using the novel low-dose stress/high-dose rest protocol will be compared to the stress/rest ratios achieved using conventional rest/stress protocols (described above). The unpaired Student's t-test will be used. In addition rest/stress count densities achieved using exercise (50 patients) and regadenoson (50 patients) with the novel protocol will be compared with stress/rest ratios achieved using standard rest/stress imaging in the exercise (59 patients) and regadenoson (29 patients) subgroups.

Primary Endpoint 1: Comparison of the myocardial count density ratio of the test group using the Rapid Protocol vs. the myocardial count density ratio of the Traditional protocol in the control group.

Secondary Endpoints

1. Image quality
2. # of patients with normal stress studies that may have had a stress-only study.
3. Reduction in radiation exposure between Test (Rapid) and Control (Traditional) groups
4. Comparison of absolute stress and rest myocardial count densities in Test and Control groups 5. Start to finish time, and potential cost savings between the two groups 6. Comparison of total radiopharmaceutical dose between the two groups

Study Duration:

1 year

Statistical Plan:

Primary endpoint: The individual stress and rest, as well as the stress:rest myocardial count density ratio will be determined from test group processed tomograms and compared with control group using UNPAIRED T TEST

Secondary: The image quality of the test group stress and rest perfusion tomograms and the gated tomograms will be graded visually using a 5-point scale: 1 (poor) - 5 (excellent), and compared with the control group using the UNPAIRED T TEST.

The overall reduction in radiation exposure to the test group will be analyzed using, as a comparator, the patient size and weight based radiopharmaceutical dose and imaging time used in a standard Stress/Rest Protocol.

The time and cost savings associated with forgoing the resting study in those patients with a normal stress scan will be calculated.

Based on a control group mean maximum contrast dose (MCD) of 4.4 and standard deviation of 9.5, this study will have greater than 80% power to detect a 0.3 difference in the MCD ratio. (Alpha=5%)

ELIGIBILITY:
Inclusion Criteria:

* adult
* not pregnant
* suspected coronary artery disease

Exclusion Criteria:

* pregnant
* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest G DePuey, M.D., Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- 'St. Luke's-Roosevelt Hospital, New York, New York, United States

REFERENCES:
- [Result] DePuey EG, Ata P, Wray R, Friedman M. Very low-activity stress/high-activity rest, single-day myocardial perfusion SPECT with a conventional sodium iodide camera and wide beam reconstruction processing. J Nucl Cardiol. 2012 Oct;19(5):931-44. doi: 10.1007/s12350-012-9596-8. Epub 2012 Jul 10. PMID 22777525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 102 consecutive patients referred for clinically indicated myocardial perfusion SPECT were recruited.
Groups:
- Stress/Rest Myocardial Perfusion SPECT Patients: All patients referred for clinically indicated myocardial perfusion SPECT are eligible candidates for this protocol. Low-dose stress/high-dose rest myocardial perfusion SPECT is performed according to the protocol and image quality and rest/stress myocardial count density ratios are assessed.
Period: Overall Study
Arm/Group | Stress/Rest Myocardial Perfusion SPECT Patients
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Myocardial Perfusion SPECT: The 102 study patients underwent a very low-activity stress/high-activity rest, single-day myocardial perfusion SPECT ith a conventional sodium iodide camera and wide beam reconstruction processing.
Arm/Group | Myocardial Perfusion SPECT
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 102
Weight [Mean (Standard Deviation); unit: pounds] | 178 (41)
Chest circumference [Mean (Standard Deviation); unit: inches] | 41.5 (4.0)
Coronary Artery Disease [Number; unit: participants] — Patients with a history of known coronary artery disease with either prior myocardial infarction, and/or coronary revascularization, and/or a history of congestive heart failure.
  participants
    yes | 53
    no | 49
Risk of Coronary Artery Disease [Number; unit: participants] — Patients presented with risk factors for coronary artery disease and symptomatology imparting an intermediate likelihood of coronary artery disease.
  participants
    yes | 37
    no | 65
Non-cardiac surgery [Number; unit: participants] — Patients had a low intermediate likelihood of coronary disease and were being evaluated pre-operatively for non-cardiac surgery.
  participants
    yes | 12
    no | 90

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Perfusion SPECT Image Quality 12 Minutes
Description: SPECT image quality realized using the stress/rest single-day protocol: 12- minute post-stress acquisitions If myocardial image quality is equivalent or superior to that encountered with standard myocardial perfusion SPECT performed using a standard low-dose rest/high-dose SPECT protocol and OSEM processing and if the rest/stress myocardial count density ratio is > 3.5 the outcome of a particular patient is judged to be favorable (acceptable).If either image quality is "poor" or if the rest/stress count density ratio is less than 3.5, the outcome is judged unfavorable.
Time Frame: at 12 minutes
Measure: Number; unit: participants
Groups:
- Myocardial Perfusion SPECT: Participants underwent novel low-dose rest/high-dose Tc-99m sestamibi SPECT protocol with wide beam reconstruction SPECT processing
Arm/Group | Myocardial Perfusion SPECT
Number analyzed (Participants) | 102
participants
  Stress non-gated Poor | 1
  Stress gated Poor | 0
  Stress non-gated Fair | 8
  Stress gated Fair | 3
  Stress non-gated Good | 30
  Stress gated Good | 20
  Stress non-gated Excellent | 63
  Stress gated | 79

2. Primary Outcome: Myocardial Perfusion SPECT Image Quality 16 Minutes
Description: SPECT image quality realized using the stress/rest single-day protocol: 16- minute post-stress acquisitions If myocardial image quality is equivalent or superior to that encountered with standard myocardial perfusion SPECT performed using a standard low-dose rest/high-dose SPECT protocol and OSEM processing and if the rest/stress myocardial count density ratio is > 3.5 the outcome of a particular patient is judged to be favorable (acceptable).If either image quality is "poor" or if the rest/stress count density ratio is less than 3.5, the outcome is judged unfavorable.
Time Frame: at 16 minutes
Population: Of the total 102 patients enrolled, additional 16-minute post-stress SPECT was performed on 37 patients.
Measure: Number; unit: participants
Arm/Group | Myocardial Perfusion SPECT
Number analyzed (Participants) | 37
participants
  Stress non-gated Poor | 0
  Stress gated Poor | 0
  Stress non-gated Fair | 1
  Stress gated Fair | 1
  Stress non-gated Good | 7
  Stress gated Good | 7
  Stress non-gated Excellent | 29
  Stress gated Excellent | 30

3. Secondary Outcome: Rest/Stress Myocardial Count Density Ratio
Description: The rest and stress myocardial count densities are determined automatically using Evolution software on the GE Healthcare Xeleris Nuclear Medicine computer workstation. The ratio is calculated by simple division.
  Please not that patient outcomes are NOT measured in this research protocol.
Time Frame: immediately following SPECT image processing (1 hour after the test)
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse Events information not collected for this study.
Arm/Group | Myocardial Perfusion SPECT
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No